CLINICAL TRIAL: NCT00279617
Title: Levetiracetam Treatment of Panic Disorder and Lactate-Induced Panic Attacks
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Lindner Center of HOPE (Other)
Collaborators: UCB Pharma (Industry); University of Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2-Miefert
Record Dates: First submitted 2006-01-18; First posted 2006-01-19 (Estimated); Last update posted 2011-12-13 (Estimated); Status verified 2011-12

CONDITIONS: Panic Disorder
MeSH Terms: conditions — Panic Disorder | interventions — Levetiracetam

ARMS (1):
- Levetricetam (Active Comparator): open label treatment
  Interventions: Drug: levetiracetam

INTERVENTIONS:
Drug: levetiracetam — open label levetricetam
  Other Names: Keppra

SUMMARY:
The main purpose of this research study is to determine whether the drug Levetiracetam (Keppra™) is effective in the prevention of panic attacks. The drug Levetiracetam (Keppra™) has been approved for the treatment of seizures by the U.S. Federal Food and Drug Administration (FDA) and is available by prescription. Levetiracetam has not been approved by the FDA for the treatment of panic disorder.

DETAILED DESCRIPTION:
a) Methods and Procedures:

Study Treatment:

Study drug and dosing: Levetiracetam open-label, with the following titration schedule to begin after the initial lactate infusion:

Study day Levetiracetam dose 1-4 250 mg 5-7 500 mg 8-10 750 mg 11-14 1000 mg 15-18 1500 mg 19-21 2000 mg 22-25 2500 mg 26-28 3000 mg 29-56 3000 mg

Levetiracetam will be titrated to maximized clinical response (total reduction of panic attacks and intervening anxiety) and minimize side effects. Subjects who develop bothersome side effects will be permitted to have a dose reduction to alleviate such side effects. Subjects unable to tolerate levetiracetam 500 mg/d will be discontinued from the trial

Study Design:

This is an 8 week open-label trial of the antiepileptic agent, levetiracetam, in the treatment of subjects who meet DSM-IV-TR criteria for panic disorder. In addition, prior to and at the conclusion of the open-label trial, subjects will participate in a 1 hour intravenous (IV) lactate infusion to determine whether levetiracetam administration blocks lactate-induced panic attacks.

Study procedures:

Screening (Visit 1): Subjects will provide written informed consent after an explanation of all study procedures. The Structured Interview for DSM-IV anxiety disorder module will be administered to confirm the diagnosis of panic disorder. A complete psychiatric and medical history will be obtained and a physical examination, including vital signs, will be performed. Subjects must experience a minimum of one panic attack per week over the month preceding the study. Inclusion/exclusion criteria will be reviewed and subjects will be assessed for compliance with these criteria. Subjects will be given a panic attack diary to record the number of panic attacks they experience each day. Subjects will be given the API. All female subjects who are able to have children will have a blood sample drawn for laboratory evaluation of β HCG. Subjects will be asked to return in one week.

Baseline (Visit 2): Subjects will return their completed panic attack diary. Subjects will then be administered the HAM-A rating scale. Vital signs will be recorded. Subjects who continue to meet inclusion/exclusion criteria will undergo the 1 hour lactate infusion.

Infusion procedure: Subjects will be recumbent in bed and made comfortable In intravenous line will be placed in the antecubital fossa and a slow intravenous infusion of 5% dextrose in water (D5W) will be administered for 28 minutes, then accelerated for 2 min. to mimic subsequent lactate infusion. The intravenous solution will be out of view of the subject behind a bedside screen. Subjects are blind to the timing of lactate administration. At time 0 (after 30 min. of D5W infusion), an infusion of 0.5 mol/L sodium DL-lactate (at body temperature) is initiated. The total dose (10 ml/kg body weight) is administered over the subsequent 20 min., unless the subject experiences a panic attack, in which case the lactate infusion is immediately discontinued. At the time of panic symptoms, or at the end of 20 min., the subject is switched back to D5W for 5 min., followed by termination of the infusion.

Subjective symptoms of a panic attack will be assessed using the 28-item Acute Panic Inventory. The API will administered at the conclusion of the screening interview during which time they will be asked to describe a typical panic attack, prior to infusion of D5W, prior to lactate infusion, halfway through lactate infusion (10 min. into the infusion), and, if precipitated, at the emergence of a panic attack. To meet criteria for having a panic attack, a subject must experience a crescendo of anxiety, fear or apprehension, and at least 4 of the physical symptoms listed in DSM-IV-TR for a panic attack. Subjects who experience a panic attack will be offered lorazepam 0.5 mg po to alleviate panic attack symptoms.

Subjects will begin open-label treatment with levetiracetam following the initial lactate infusion. Levetiracetam will be titrated according to the schedule described above.

Subjects who do not experience a lactate induced panic attack at baseline will be eliminated from the study.

Day 7 (Visit 3): The HAM-A will be administered and panic attack diaries will be reviewed and recorded. Adverse events will be reviewed. Vital signs will be recorded. Study medication will be reviewed for adherence. Study medication will be dispensed.

Day 14 (Visit 4): The HAM-A will be administered and panic attack diaries will be reviewed and recorded. Adverse events will be reviewed. Vital signs will be recorded. Study medication will be reviewed for adherence. Study medication will be dispensed.

Day 28 (Visit 5): The HAM-A will be administered and panic attack diaries will be reviewed and recorded. Adverse events will be reviewed. Vital signs will be recorded. Study medication will be reviewed for adherence. Study medication will be dispensed.

Day 42 (Visit 6): The HAM-A will be administered and panic attack diaries will be reviewed and recorded. Adverse events will be reviewed. Vital signs will be recorded. Study medication will be reviewed for adherence. Study medication will be dispensed.

Day 56 (Visit 7): The HAM-A will be administered and panic attack diaries will be reviewed and recorded. Adverse events will be reviewed. Vital signs will be recorded.

Subjects will repeat the lactate infusion procedure as described in Visit 2. At the conclusion of the second lactated infusion, subjects who have responded to treatment with levetiracetam will be offered up to 3 months continued treatment with levetiracetam and office visits at no charge until subjects are appropriately referred for continued follow-up treatment. Subjects not responding to levetiracetam treatment will be offered treatment with an FDA-approved medication for panic disorder.

ELIGIBILITY:
Inclusion Criteria:

1. Outpatient subjects age 18 years or older.
2. Subjects must meet DSM-IV-TR criteria for panic disorder with or without agoraphobia.
3. Subjects must experience a minimum of one panic attack per week over the month preceding the study.
4. Subjects must be fluent in English.
5. Subjects must be able to provide and understand written informed consent.

Exclusion Criteria:

1. Subjects unable to provide and understand written informed consent.
2. Subjects previously treated with levetiracetam.
3. Subjects who meet DVM-IV-TR criteria for current diagnosis of mood, psychotic or substance use disorder.
4. Subjects who have acute or unstable medical illness.
5. Subjects with a history of seizures or structural brain damage from trauma.
6. Subjects currently receiving successful treatment for panic disorder (i.e., subjects will not have medications discontinued to participate in the study if they are effective in the treatment of their panic attacks).
7. Subjects susceptible to lactate infusions.
8. Female subjects who are pregnant or lactating.
9. Female subjects who, if fertile, are not using medically acceptable and reliable method of contraception.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2006-01; Primary Completion 2009-02 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Hamilton Anxiety scale (HAM-A) | each visit

CONTACTS AND LOCATIONS:
Overall Officials: Paul Keck, MD, Principal Investigator — University of Cincinnati
Locations (1):
- University of Cincinnati Medical Center, Cincinnati, Ohio, United States